CLINICAL TRIAL: NCT02160912
Title: Non Interventional Study Regarding the Application of Ectoin Mund- & Rachenspray in Patients With Acute Laryngitis and/or Acute Pharyngitis
Brief Title: Non Interventional Study (NIS) Regarding the Application of Ectoin Mund- & Rachenspray in Patients With Acute Laryngitis and/or Acute Pharyngitis
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: EctMRS/aLR/2014
Record Dates: First submitted 2014-06-04; First posted 2014-06-11 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Acute Pharyngitis; Acute Laryngitis
MeSH Terms: conditions — Croup

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ectoin Mund- & Rachenspray: treatment with Ectoin Mund- & Rachenspray 1%
- Emser Pastillen: treatment with Emser Pastillen

SUMMARY:
In this observational study insights regarding the tolerability and influence on the quality of life of the topical treatment Ectoin Mund- and Rachenspray compared to Emser Pastillen in patients with acute Pharyngitis/ Laryngitis under real life conditions shall be gained.

Patients are treated with Ectoin Mund- & Rachenspray 1% or Emser Pastillen according to the demands of the physician and the instructions for use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute Laryngitis and/or Pharyngitis which are already treated with Ectoin Mund- & Rachenspray 1% or Emser Pastillen

Exclusion Criteria:

* contraindications according to instructions for use

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care unit In this non interventional study the therapy process of a total of 90 patients with acute pharyngitis and/or laryngitis for which the physician has planned a therapy with Ectoin Mund- & Rachenspray 1% (60 Patients) or Emser Pastillen (30 patients) shall be observed in 8 clinical centers
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Pharyngitis symptom score evaluated by the physician | Visit 1, Visit 2 (after 3 days), Visite 3 (after 7 days)
  Assessment of the symptoms of pharyngitis on a 4 point scale (none, mild, moderate strong):
  * swollen palatine tonsils
  * swollen lymph nodes in the throat
  * fever
  * cough

SECONDARY OUTCOMES:
Change in patient's general condition evaluated by the physician | Visit 1, Visit 2 (after 3 days), Visit 3 (after 7 days)
  Physician's assessment of the general conditions on a 4 point scale (good condition, slightly reduced condition, bad condition, very bad condition)
Change in Evaluation of the hoarseness | Visit 1, Visit 2 (after 3 days), Visit 3 (after 7 days)
  physician's assessment of the hoarseness of the patient on a 4 point scale (none, mild, moderate, strong)
Change in Dysphagia | Visit 1, Visit 2 (after 3 days), Visit 3 (after 7 days)
  physician's assessment of dysphagia of the patient on a 4 point scale (none, mild, moderate, strong)
Change in efficacy evaluation by the physician | Visit 1, Visit 2 (after 3 days), Visit 3 (after 1 week)
  Assessment of the efficacy on a 4 point scale (0= bad, 1=sufficient, 2=good, 3=very good)
Change in efficacy evaluation by the patient | Visit 1, Visit 2 (after 3 days), Visit 3 (after 7 days)
  Assessment of the efficacy on a 4 point scale (0_bad, 1=sufficient, 2=good, 3=very good)
Change in Evaluation of the tolerability by the physician | Visit 1, Visit 2 (after 3 days), Visit 3 (after 7 days))
  Assessment of the tolerability by the physician on a 4 point scale (0= bad, 1=sufficient, 2=good, 3=very good)
Change in Evaluation of the tolerability by the patient | Visit 1, Visit 2 (after 3 days), Visit 3 (after 7 days))
  Assessment of the tolerability by the patient on a 4 point scale (0= bad, 1=sufficient, 2=good, 3=very good)
Change in number and type of adverse events | Visit 2 (after 3 days) Visit 3 (after 7 days)
  incidence of adverse events and correlation with the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mösges, MD, Principal Investigator — Klinikum der Universität zu Köln
Locations (8):
- Germany (8):
  - Norbert Pasch-Facharzt für HNO Heilkunde, Aachen
  - HNO Praxis Aachen Brand, Aachen
  - Taufik Shahab -Facharzt für HNO Heilkunde, Cologne
  - Bey - Facharzt f. HNO Heilkunde, Cologne
  - HNO-Praxis Peter Hinterkausen & Dr. med. Eva Bottler-Neufert, Cologne
  - HNo Praxis Dr. Uta Thieme, Duisburg
  - Dr. Lenzenhuber-Fachärztin für HNO Heilkunde, Jülich
  - Wilhelm Schütz -Facharzt für HNO Heilkunde, Jülich